CLINICAL TRIAL: NCT01223053
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Parallel-Group, Confirmatory Phase 3 Study to Assess the Efficacy and Safety of TDLP-110 (Ketotransdel®, Ketoprofen 10% Cream) in the Treatment of Pain Associated With Mild to Moderate Acute Soft Tissue Injury
Brief Title: Ketoprofen 10% Cream for Treatment of Pain Associated With Mild to Moderate Acute Soft Tissue Injury
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Revised Development Program
Sponsor: Imprimis Pharmaceuticals, Inc. (Industry)
Responsible Party: Joachim Schupp, M.D., Transdel Pharmaceuticals, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDLP-110-002
Record Dates: First submitted 2010-10-08; First posted 2010-10-18 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Sprain
Keywords: Sprain; Strain; Pain; Ankle Pain; Knee Pain; Wrist Pain; Hand Pain
MeSH Terms: conditions — Sprains and Strains; Pain | interventions — Ketoprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Active (Active Comparator): Topical ketoprofen 10% Cream
  Interventions: Drug: Ketoprofen 10% cream
- Placebo Cream (Placebo Comparator): Placebo Cream
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketoprofen 10% cream — 100 mg (10%) in 1 gram of topical cream applied three times per day for 7 days. Safety follow up on day 14.
  Other Names: TDLP-110, Ketotransdel
  Arms: Active
Drug: Placebo — Matching placebo cream containing identical constituents as the active comparator except for ketoprofen
  Arms: Placebo Cream

SUMMARY:
Transdel Pharmaceuticals is investigating a topical cream formulation consisting of 10% ketoprofen for the local treatment of pain associated with mild to moderate acute soft tissue injury in this confirmatory Phase 3 trial.

DETAILED DESCRIPTION:
This Phase 3 study examines the use of TDLP-110 (a.k.a. Ketotransdel® or ketoprofen 10% cream), as a topical treatment for pain associated with mild to moderate acute soft tissue injury of the upper and lower extremities to serve as a confirmatory trial. The first completed Phase 3 study showed efficacy and safety of TDLP-110 compared to placebo in improving the patient assessment of pain.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female and 18 to 75 years of age, inclusive.
* Female patients of childbearing potential must practice abstinence or be using a medically acceptable form of contraception
* Have a diagnosis of uncomplicated acute soft tissue injury of the upper or lower extremity, including acute injuries of ligaments, tendons, or muscles (including Grade 1 or Grade 2 sprain or strain), that has occurred within the 60 hours preceding the baseline visit.
* Meet pain intensity criteria
* Are willing to discontinue use of any pain medication or treatments not provided as part of the study.

Exclusion Criteria:

* Participation in a previous clinical study with the drug TDLP-110 (ketoprofen 10% cream).
* Are pregnant or lactating.
* Have a Grade 3 sprain or strain, bilateral sprain or strain, or concomitant fracture or open wound at the site of the sprain or strain, or have a serious injury, as determined by the investigator
* Have a shoulder (rotator cuff) injury.
* Have been treated for a sprain or strain of the same site within the past 3 months.
* Have contusions at the site of acute soft tissue injury intended for treatment.
* Have active skin lesions or disease at the intended site of application of the study medication.
* Have had pharmacologic treatment for the injury less than 24 hours before the baseline assessments
* Use of any oral or parenteral corticosteroids within 30 days of injury.
* Have had non-pharmacologic treatments of the injury other than rest, ice, compression, and/or elevation (RICE) within 12 hours prior to the baseline visit.
* Have a history or physical examination finding that is incompatible with safe participation in the study.
* Have a history or physical examination finding that is, in the opinion of the investigator, incompatible with study product use or with obtaining interpretable data.
* Are taking medications or other substances contraindicated due to the nature of the study medication or with the potential for drug interactions.
* Are allergic or sensitive to soy lecithin or soy lecithin-containing products.
* Are taking probenecid or similar drugs that may significantly affect renal function.
* Are taking a sleep medication, sedative hypnotic, anxiolytic, or antidepressant medication at a dose that has not been stable for at least 2 months.
* Are receiving physical therapy for the index injury
* Have scheduled elective surgery or other invasive procedures during the period of study participation.
* Have any illness or concurrent condition that would, in the opinion of the investigator, make study participation unsafe or would confound study results ly undergoing treatment for chronic pain, or severe systemic disease).
* Have received an investigational drug or product or participated in an investigational drug study within a period of 30 days prior to receiving study medication.
* Have an active worker's compensation claim or personal injury claim regarding injury to the index site.
* Are suspected by the investigator of recent or current drug or alcohol abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean pain intensity (100 mm VAS) during daily activities over the past 24 hours at the Day 3 visit (Day 3 +1) | 3 days

SECONDARY OUTCOMES:
CPRA; Pain curves over time; Percent change from baseline | 7 days
  * Cumulative proportion of responders for the change from baseline in mean pain intensity as assessed on the 100-mm VAS during daily activities over the past 24 hours at Day 3.
  * Change from baseline in three-times-daily pain intensity using VAS ratings recorded in the patient diaries over 7 days of treatment.
  * Percent change from baseline in pain intensity during daily activities over the past 24 hours at Day 3